CLINICAL TRIAL: NCT06968260
Title: Comparing Physiological Stress and Learning Outcomes in Instructor- vs. Software-Guided VR Basic Life Support Training
Brief Title: Stress and Learning in Educator- vs. Software-Guided VR Training for Basic Life Support
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Acibadem University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2024-17/647
Record Dates: First submitted 2025-04-28; First posted 2025-05-13 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-05

CONDITIONS: Machine Guidance; Instructor Guidance

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Machine Guidance (Experimental): The participants will receive a machine guided education
  Interventions: Other: Education Type
- Instructor Guidance (Experimental): Participants will receive human guided education
  Interventions: Other: Education Type

INTERVENTIONS:
Other: Education Type — Machine Guidance group will receive education from a software, while the Instructor Guidance Group will receive education from a human instructor.

SUMMARY:
This randomized controlled trial will explore how instructor type-human vs. machine-affects performance, immersion, and stress during VR-based Basic Life Support (BLS) training. Participants will receive VR based education wither with a machine instructor or a human instructor and complete a simulated emergency exam. Outcomes will include procedural accuracy, physiological stress (measured via electrodermal activity), and subjective evaluations of presence and instructor effectiveness.

DETAILED DESCRIPTION:
In high-stakes medical emergencies, both technical proficiency and psychological resilience are critical. Traditional Basic Life Support (BLS) training methods-such as lectures, role-play, and manikin-based practice-help students build core skills but often fall short in replicating the stress and complexity of real-world crises. As medical education evolves, virtual reality (VR) is emerging as a promising tool, offering immersive, controlled environments that simulate emergency conditions while supporting both skill acquisition and psychological engagement. However, while VR's benefits for technical training are well-established, its impact on stress management and mental preparedness remains underexplored.

This study will examine how the type of instructor-human or machine-within a VR-based training environment influences students' performance, immersion, and stress responses during BLS training. Participants will undergo VR-based BLS instruction led by either a human educator or a software-based guide, followed by a simulated emergency exam. Outcomes will be assessed through procedural accuracy, physiological stress measured via electrodermal activity (EDA), and subjective evaluations of presence and instructor effectiveness.

The findings are expected to shed light on how different instructional approaches in VR affect not only learning outcomes but also students' capacity to manage stress in high-pressure situations. By identifying how instructor type influences both competence and psychological resilience, this research aims to optimize VR-based medical training for the demands of real-world clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Being older than 18

Exclusion Criteria:

* prior completion of Basic Life Support (BLS) training
* history of virtual reality (VR)-induced motion sickness
* medical conditions such as vertigo or the use of medications known to cause vertigo-like symptoms

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 66 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Electrodermal Activity | Up to 4 weeks
  Electrodermal activity will be used to operationalize stress levels via Shimmer3 GSR+ (Galvanic Skin Response) Unit.
Presence Levels | Up to 4 weeks
  Presence will be measured using Presence Questionnaire. The questionnaire is 7- point likert type, with higher scores meaning increased presence. The minimum possible score is 1 and the maximum is 7.
Instructional Skills Questionnaire | Up to 4 weeks
  This questionnaire will be used to assess instructor evaluations. Items are rated on a 7-point Likert scale. Higher scores indicate better satisfaction with the course.
Exam Scores | Up to 4 weeks
  Scores on the exam module will be compared across groups. Scores will range from 1 to 100. Higher scores will indicate higher success.